CLINICAL TRIAL: NCT00519428
Title: Combining Antidepressants to Hasten Remission From Depression
Brief Title: Does Dual Therapy Hasten Antidepressant Response?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: University of Ottawa (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5476; 5R01MH076961-04 (NIH)
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
Keywords: depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- escitalopram + bupropion (Experimental): escitalopram plus bupropion extra long (XL) as dual treatment (i.e., this is not a SINGLE treatment arm; all patients assigned this arm received both medications)
  Interventions: Drug: escitalopram + bupropion
- escitalopram (Active Comparator): escitalopram monotherapy
  Interventions: Drug: escitalopram
- bupropion (Active Comparator): bupropion extra long (XL) monotherapy
  Interventions: Drug: bupropion extra long (XL)

INTERVENTIONS:
Drug: escitalopram — 10mg/d increasing by 10 mg/week to a maximum of 40 mg/d if tolerated and not remitted
  Other Names: Lexapro
  Arms: escitalopram
Drug: bupropion extra long (XL) — 150mg/d increasing to 300 mg/d after 1 week and 450 mg/d after 3 weeks, all increases if tolerated and not remitted
  Other Names: Wellbutrin extra long (XL)
  Arms: bupropion
Drug: escitalopram + bupropion — same dosing schedule as for monotherapy
  Other Names: Lexapro; Wellbutrin
  Arms: escitalopram + bupropion

SUMMARY:
This study will utilize a randomized double-blind design to evaluate whether initial treatment with two anti-depressant medications (escitalopram and bupropion) results in more rapid remission and greater over-all remission rates than either monotherapy in 240 depressed subjects.

DETAILED DESCRIPTION:
Depression is a major public health problem due to its prevalence and accompanying dysfunction and costs. Depression is undertreated, but even when treatment is adequate and effective, sources of delay in current pharmacologic strategies include: mechanistic delays, those related to the physiologic and behavioral effects of antidepressants; dosing delays in identifying the effective dose; and programmatic delays in identifying an effective agent using sequential monotherapy. This study will randomize 240 patients with Diagnostic and Statistical Manual, 4th Edition (DSM-IV) Major Depressive Disorder (MDD) to 12 week double blind treatment with combined escitalopram and bupropion or each antidepressant administered alone to evaluate whether combined escitalopram and bupropion result in more rapid remission and greater over-all remission than monotherapy. Preclinical and clinical studies suggest that bupropion might prevent one mechanistic delay inherent in escitalopram monotherapy. Rapid dose escalation may counter dosing delays. The simultaneous use of two known antidepressant medications may alleviate programmatic delays inherent in usual sequential monotherapy. Six months follow up and careful assessment of adverse events will address tolerability, acceptability, sustainability, and pharmacoeconomic concerns. If successful, this study might have a significant impact on clinical practice, public health, and depression's cost consequences.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18-65
2. Major Depressive Disorder as primary diagnosis
3. Physically healthy
4. Signs informed consent
5. Montgomery Asberg Depression Rating Scale (MADRS) >= 22

Exclusion Criteria:

1. Bipolar Disorder (ie, Bipolar I, Bipolar II, Bipolar NOS)
2. Life-time history of psychosis
3. Current (ie, last 6 months) drug or alcohol abuse or dependence (except nicotine)
4. Currently taking effective antidepressant medication
5. Prior adequate treatment in current depressive episode with a selective serotonin re-uptake inhibitor (SSRI), bupropion (BUP) or bupropion (BUP) + a selective serotonin re-uptake inhibitor (SSRI) ("adequate" is defined as >= 4 weeks taking >= 2/3 Physician's Desk Reference (PDR) maximal dose
6. Most recent antidepressant was within 5 weeks for fluoxetine and 1 week for all others
7. Currently taking a medication contraindicated with either study medication
8. Life time history of anorexia or bulimia
9. Life time history of seizure or known increased seizure risk (e.g., history of significant brain trauma, taking pro-convulsant medication, known anatomical brain lesion)
10. Currently taking psychoactive medication deemed to be necessary (including but not limited anticonvulsants, antidepressants, antipsychotics, steroids, and B-blockers); occasional use of hypnotics (ie, less than three times per week) will be allowed
11. Unstable medical condition (ie, condition not adequately stabilized for >= 3 months)
12. Prior intolerance to escitalopram (ESC) or bupropion (BUP)
13. Inadequate understanding of English (for US site; Canadian site permits French fluency)
14. Currently pregnant or breast-feeding; fecund women not using adequate contraceptive methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2007-08; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, M.D., Principal Investigator — New York State Psychiatric Institute; Pierre Blier, M.D., Principal Investigator — University of Ottawa
Locations (2):
- New York State Psychiatric Institute, New York, New York, United States
- University of Ottawa, Institute of Mental Health Research, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Wijk G, Enkhbold Y, Cnudde K, Szostakiwskyj MW, Blier P, Knott V, Jaworska N, Protzner AB. One size does not fit all: notable individual variation in brain activity correlates of antidepressant treatment response. Front Psychiatry. 2024 Apr 2;15:1358018. doi: 10.3389/fpsyt.2024.1358018. eCollection 2024. PMID 38628260
- [Derived] Weissman MM, Wickramaratne P, Pilowsky DJ, Poh E, Batten LA, Hernandez M, Flament MF, Stewart JA, McGrath P, Blier P, Stewart JW. Treatment of maternal depression in a medication clinical trial and its effect on children. Am J Psychiatry. 2015 May;172(5):450-9. doi: 10.1176/appi.ajp.2014.13121679. Epub 2015 Jan 23. PMID 25615566
- [Derived] Gerra ML, Marchesi C, Amat JA, Blier P, Hellerstein DJ, Stewart JW. Does negative affectivity predict differential response to an SSRI versus a non-SSRI antidepressant? J Clin Psychiatry. 2014 Sep;75(9):e939-44. doi: 10.4088/JCP.14m09025. PMID 25295437
- [Derived] Stewart JW, McGrath PJ, Blondeau C, Deliyannides DA, Hellerstein D, Norris S, Amat J, Pilowsky DJ, Tessier P, Laberge L, O'Shea D, Chen Y, Withers A, Bergeron R, Blier P. Combination antidepressant therapy for major depressive disorder: speed and probability of remission. J Psychiatr Res. 2014 May;52:7-14. doi: 10.1016/j.jpsychires.2013.12.001. Epub 2013 Dec 17. PMID 24485847
- See also: Depression Evaluation Service official website — http://depression-nyc.org/
- See also: Columbia University Depart,ment of Psychiatry web page — https://www.columbiapsychiatry.org/
- See also: official website of the University of Ottawa's Institute of Mental Health Research — http://www.imhr.ca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: August, 2007 to August 2011 Locations: 4 outpatient research clinics in two countries (US and Canada)
Pre-assignment Details: All patients had to be psychoactive drug-free for at least two weeks (five weeks for fluoxetine) prior to randomization and had to continue to meet study entry criteria at point of randomization
Groups:
- Escitalopram + Bupropion: escitalopram plus bupropion
- Bupropion: bupropion monotherapy
Period: Overall Study
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Started | 78 | 84 | 83
Completed | 57 | 69 | 58
Not Completed | 21 | 15 | 25
Not completed — Adverse Event | 5 | 2 | 10
Not completed — Lost to Follow-up | 7 | 7 | 6
Not completed — Withdrawal by Subject | 8 | 3 | 7
Not completed — unstated | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Escitalopram + Bupropion: escitalopram plus bupropion XL
- Bupropion: bupropion XL monotherapy
- Total: Total of all reporting groups
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion | Total
Number analyzed (Participants) | 78 | 84 | 83 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient's report of their age
  years
    Age | 40 (10) | 41 (11) | 40 (11) | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 62 | 49 | 163
  Male | 26 | 22 | 34 | 82
Region of Enrollment [Number; unit: participants]
  United States | 37 | 42 | 41 | 120
  Canada | 41 | 42 | 42 | 125

OUTCOME MEASURES:

1. Primary Outcome: Time to Remission, Defined by the Week of Onset of Persistent Hamilton Rating Scale for Depression (HAM-D 17) <= 7, With no Subsequent HAM-D 17 > 7
Description: Life Table Survival Analysis run twice, once comparing Dual Therapy (i.e., Bupropion + Escitalopram) to Bupropion alone (i.e., Bupropion + Placebo) and once comparing Dual Therapy to Escitalopram alone (i.e., Escitalopram + Placebo). Because both analyses must significantly favor Dual Therapy, each individual analysis must reach a critical alpha = .0916 in order to reach an over-all alpha = .05.
Time Frame: 12 weeks
Population: age 18-65 with Major Depressive Disorder (MDD), non-bipolar, non-psychotic, non-substance abusing, without intolerance to study drugs or adequate selective serotonin re-uptake inhibitor (SSRI) and/or bupropion treatment in current episode; physically healthy without contraindications to bupropion or escitalopram.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Number analyzed (Participants) | 78 | 84 | 83
weeks | 8 (7) | 9 (7) | 10 (7)
Statistical Analysis 1: Comparison: Escitalopram + Bupropion vs Escitalopram vs Bupropion; Hypothesis: Dual Treatment (escitalopram + bupropion) will result in greater improvement over 12 weeks than either monotherapy (i.e., two analyses: 1) dual treatment will outperform escitalopram monotherapy; 2) dual treatment will outperform bupropion monotherapy). Therefore each analysis will be done twice and it will be required that both analyses be significant to declare the over-all study significant; Test type: Superiority — Hypothesis: Dual Treatment (escitalopram + bupropion) will result in greater improvement over 12 weeks than either monotherapy (i.e., two analyses: 1) dual treatment will outperform escitalopram monotherapy; 2) dual treatment will outperform bupropion monotherapy); p = .05, Cochran-Mantel-Haenszel — Each individual test will require the calculated "p" to be < .0916 to declare that comparison to be significant. Since the hypothesis requires both comparisons to be significant, this produces an over-all alpha of .05; Mean Difference (Final Values) = .05, Standard Deviation 4

2. Secondary Outcome: Remission: Persistent Hamilton Rating Scale for Depression, 17 Items (HAM-D 17) <= 7, With no HAM-D 17 >7 Through Week 12
Description: Chi square comparison of rates of persistent remission (i.e., no subsequent Hamilton Rating Scale for Depression, 17 items [HAMD-D 17] > 7 once HAMD-D 17 <= 7); Dual rate vs. Escitalopram only rate and Dual rate vs. Bupropion only rate.
Time Frame: 12 weeks
Population: age 18-65 with MDD, non-bipolar, non-psychotic, non-substance abusing, without intolerance to study drugs or adequate SSRI/bupropion treatment in current episode; physically healthy without contraindications to bupropion or escitalopram.
Measure: Number; unit: percentage of participants
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Number analyzed (Participants) | 78 | 84 | 83
percentage of participants | 52 | 46 | 34

3. Secondary Outcome: Severity of Depressive Symptoms as Measured by Hamilton Rating Scale for Depression (HAM-D 17)
Description: Last summary score rating on the 17-item Hamilton Rating Scale for Depression Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. Range 0-58.
  0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on Hamilton Rating Scale for Depre
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Number analyzed (Participants) | 78 | 83 | 84
units on Hamilton Rating Scale for Depre | 10 (8) | 9 (7) | 12 (8)
Statistical Analysis 1: Comparison: Escitalopram + Bupropion vs Escitalopram vs Bupropion; To test the hypothesis that escitalopram + bupropion would have superior efficacy relative to each monotherapy, the group receiving both medications was separately compared to each monotherapy group, covarying for baseline score and country; Test type: Superiority or Other; p = .0916, ANCOVA — escitalopram + bupropion vs. escitalopram: F(1,159) = 1.93, ns escitalopram + bupropion vs. bupropion: F (1,157) = 1.99, ns; adjusting for baseline score and country; Mean Difference (Final Values) = 10, Standard Deviation 8

4. Secondary Outcome: Functioning, as Measured by the Social Adjustment Scale (SAS) Summary Score
Description: Social adjustment was measured using the Social Adjustment Scale (SAS). The SAS is a self-report scale that assesses depressive symptoms and functioning in nine social and work-related domains generating a total score that is indicative of a subject's overall level of social adjustment. Subjects rate their own social functioning over times on a 5-point scale on items covering work for pay, housework, extended family, parenting, marital status, social activity and leisure, family unit and student status (sub-scales). Mean values of all the sub-scales are used, with a range from 0-5. Higher score = worse outcome … worse functioning
Time Frame: 12 weeks
Population: All randomized patients; latest available Total SAS score used if week 12 score not available.
Measure: Mean (Standard Deviation); unit: units on the SAS scale
Groups:
- Escitalopram + Bupropion: escitalopram plus bupropion XL as dual treatment (i.e., this is not a SINGLE treatment arm; all patients assigned this arm received both medications)
  escitalopram + bupropion: same dosing schedule as for monotherapy
- Bupropion: bupropion XL monotherapy
  bupropion XL: 150mg/d increasing to 300 mg/d after 1 week and 450 mg/d after 3 weeks, all increases if tolerated and not remitted
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Number analyzed (Participants) | 78 | 83 | 84
units on the SAS scale | 2.65 (.69) | 2.63 (.69) | 2.74 (.71)

5. Secondary Outcome: Quality of Life, as Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Short Form (SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) intends to measure quality of life in 16 domains. A summary score is computed by adding the scores and dividing by 16 (or the number of answered items if some are not answered).
  The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70. Higher score means more satisfaction.
Time Frame: 12 weeks
Population: All Randomized Subjects
Measure: Mean (Standard Deviation); unit: units on the Q-LES-Q scale
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Number analyzed (Participants) | 78 | 83 | 84
units on the Q-LES-Q scale | 3.0 (.82) | 3.0 (.76) | 3.1 (.74)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: A modified Systematic Assessment for Treatment Emergent Events (SAFTEE) at each visit specifically asked about 17 items (too much energy, muscle tightness, insomnia, tremor, poor concentration, word finding, spacy, dizzy, headache, dry mouth, decreased appetite, nausea, low energy, sleepy, sweating, decreased libido, anger/irritability) a pilot study showed occurred in at least 10% of patients treated with escitalopram plus bupropion. A General Inquiry then asked re additional symptoms.
Arm/Group | Escitalopram + Bupropion | Escitalopram | Bupropion
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/84 | 0/83
Other Adverse Events (participants affected / at risk) | 71/78 | 80/84 | 71/83
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram + Bupropion (N=78) | Escitalopram (N=84) | Bupropion (N=83)
Too much energy (General disorders) | 5 (5) | 4 (4) | 7 (7) — A feeling of being too "revved up"
muscle tightness (Musculoskeletal and connective tissue disorders) | 13 (13) | 14 (14) | 18 (18) — a feeling of tenseness or tightness in the muscles
insomnia (General disorders) | 24 (24) | 27 (27) | 31 (31) — trouble falling asleep, staying asleep or waking too early
tremor (Nervous system disorders) | 23 (23) | 14 (14) | 18 (18) — involuntary shaking or trembling
trouble thinking (Nervous system disorders) | 12 (12) | 13 (13) | 5 (5) — trouble thinking or concentrating, cognitive disturbance
trouble finding words (Nervous system disorders) | 5 (5) | 6 (6) | 7 (7) — word finding difficulty
spacey (Nervous system disorders) | 13 (13) | 12 (12) | 5 (5) — feeling "spacey", "out of it", "fuzzy headed", "cotton in my head"
dizzy (Cardiac disorders) | 19 (19) | 20 (20) | 19 (19) — feeling dizzy, lightheaded or faint
headache (Nervous system disorders) | 28 (28) | 28 (28) | 26 (26) — pain inside the head
dry mouth (Gastrointestinal disorders) | 27 (27) | 18 (18) | 28 (28) — dry mouth
decreased appetite (Gastrointestinal disorders) | 17 (17) | 21 (21) | 21 (21) — anorexia
nausea, vomiting (Gastrointestinal disorders) | 25 (25) | 32 (32) | 28 (28) — nausea, vomiting, queasy stomach
lethargy (General disorders) | 10 (10) | 15 (15) | 10 (10) — low energy, lack of "get up and go"
daytime sleepiness (Nervous system disorders) | 13 (13) | 17 (17) | 9 (9) — daytime sleepiness, feeling sleepy or groggy during the day
sweating (General disorders) | 19 (19) | 13 (13) | 5 (5) — sweating too much, excessive perspiration
sexual dysfunction (General disorders) | 20 (20) | 18 (28) | 9 (9) — delayed orgasm, anorgasmia, erectile dysfunction, poor libido, low sex drive
anger, irritability (Psychiatric disorders) | 4 (4) | 5 (5) | 14 (14) — anger, irritability, feeling like "flying off the handle", too touchy

LIMITATIONS AND CAVEATS:
Sample size may have limited demonstration of differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No